CLINICAL TRIAL: NCT04380272
Title: Development of an Assessment Method for Obstructive Tonsillar Hypertrophy in Children by Ultrasonography (Pamukkale Technique)
Brief Title: Development of an Assessment Method for Obstructive Tonsillar Hypertrophy in Children by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erdem Mengi, Assistant Professor of Otorhinolaryngology, Pamukkale University
Other Study IDs: 60116787-020/81401
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Obstructive Tonsillar Hypertrophy
Keywords: tonsil; tonsillar hypertrophy; ultrasonography; children

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brodsky tonsil staging system: An oropharynx examination of all participants will be performed and tonsil size will be evaluated according to the Brodsky staging system. According to this staging system, tonsil sizes will be classified as stage I when the tonsils fill less than 25% of the transverse oropharyngeal space measured between the anterior tonsillar pillars; stage II when they fill between 25% and 50%, stage III when they fill between 50% and 75%, and stage IV when they fill more than 75%.
- The ultrasonographic data: The submental ultrasonography will be performed on all participants. Ultrasonographic examinations will be performed blinded to the physical examination results. All measurements will be performed by the same radiologist with experience in the field of ultrasonography. A GE LOGIQ E9 (GE Healthcare, Milwaukee, WI, USA) device will be used in the ultrasonography examination. The participants will be viewed using a 2-9 MHz linear probe from the submental region. The examination will be performed while the patient was lying in a supine position with a support placed under the neck.
  Interventions: Diagnostic Test: The ROC analysis

INTERVENTIONS:
Diagnostic Test: The ROC analysis — The Brodsky clinical stage and ultrasonographic data of the participants will be matched, and the diagnostic value of the submental US in the classification of tonsil hypertrophy as non-obstructive and obstructive will be evaluated. A ROC analysis will be used to determine the optimal cut-off value.
  Groups: The ultrasonographic data

SUMMARY:
Chronic tonsillar hypertrophy is one of the most common causes of upper airway obstruction in children. Currently, several clinical staging systems are used to evaluate airway obstruction due to tonsillar hypertrophy. However, as these staging systems are based on a physical examination, it is not always possible to accurately evaluate the tonsil size, especially in children, and so objective and reliable methods are required in this field. In this study, the investigators aimed to develop a new method for the objective evaluation of airway obstruction due to tonsillar hypertrophy using submental ultrasonography (US) in children.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most frequently performed operations in childhood, and one of the most important indications of this surgery is chronic tonsillar hypertrophy. Chronic tonsillar hypertrophy accounts for 80% of cases with obstructive sleep apnea syndrome (OSAS) in childhood, and growth and development delay, low academic performance, facial developmental abnormalities, and cardiopulmonary diseases may emerge as a result. For this reason, an accurate evaluation of tonsil size is crucial both during clinical follow-up and in tonsillectomy decisions.

Currently, several clinical staging systems are used to evaluate tonsil size in children, with the "Brodsky" and "Friedman" scales being the most commonly used systems. These staging systems make use of a physical examination, with tonsil hypertrophies generally classified into 4 stages based on the extension of the tonsil from the anterior plica to the midline. Stages 3 and 4 tonsil hypertrophy are generally accepted as obstructive, and a tonsillectomy decision is made when clinical complaints support this. For such an evaluation of tonsil grade, the child should be cooperative, should easily open his/her mouth, and should not gag. In the event of the patient's non-compliance, the size of the tongue and tongue base, the hyperactive gag reflex, and trismus may challenge this evaluation. The gag reflex during the examination causes the tonsils to move towards the midline, making the tonsils seem bigger than the real size. An obstruction at the hypopharyngeal level due to hypertrophic tonsils may be missed due to poor visualization of the inferior pole of the tonsil in patients with a large tongue. For these reasons, a correct clinical evaluation of the tonsil size may not always be possible through a physical examination. Thus objective and reliable methods are required for the classification of tonsillar hypertrophy.

There have been no studies to date investigating the use of ultrasonography (US) in the evaluation of airway obstruction due to tonsillar hypertrophy, despite the advantages of high patient compliance, low cost, and no radiation exposure. The present study suggests a new method for the evaluation of airway obstruction due to tonsillar hypertrophy using the submental US in children.

ELIGIBILITY:
Inclusion Criteria:

* The pediatric patients

Exclusion Criteria:

* Adult patients
* Patients identified with active infections

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The pediatric patients who presented to the otorhinolaryngology outpatient clinic with complaints of recurrent tonsillitis, snoring, and/or witnessed apnea between January 2019 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of tonsil size according to the Brodsky tonsil staging system | 20 minutes
  The investigators will classify the Brodsky Stage I and II cases as non-obstructive tonsillar hypertrophy and the Brodsky stage III and IV as obstructive tonsillar hypertrophy.
The ultrasonographic intertonsillar distance, transverse length of the tongue base and the ratio of intertonsillar distance/transverse length of the tongue base | 20 minutes
  After the neck of the participant will be brought to extension, the ultrasound probe will be placed on the submental region, and both tonsils will be visualized in the midline in the transverse plane. The narrowest airway space will be marked between the two tonsils and the intertonsillar distance (ITD) will be measured. Subsequently, in the same region, the attachments of the palatoglossal muscles to the tongue base, as the projection of the anterior plicae, will be determined, and the widest transverse length of the tongue base (TLTB) at this level will be measured. The ratio of ITD to TLTB will be calculated for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Mengi, Principal Investigator — Pamukkale Üniversitesi Tıp Fakültesi
Locations (1):
- Erdem Mengi, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No